CLINICAL TRIAL: NCT01702857
Title: A Phase I, Randomized, Placebo-Controlled, Observer-blind, Two-dose (0-28 Day Schedule) Primary Vaccination Study of WRAIR Tetravalent Dengue Virus Purified Inactivated Vaccine (TDENV-PIV) in Healthy Adults in Puerto Rico
Brief Title: A Two-dose Primary Vaccination Study of a Tetravalent Dengue Virus Purified Inactivated Vaccine vs. Placebo in Healthy Adults (in Puerto Rico)
Acronym: DPIV-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S-12-12; 116614 (Other: GSK); WRAIR 1945 (Other: WRAIR); DPIV-002 (Other: GSK Protocol #)
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Dengue Fever
Keywords: Dengue; Dengue fever; Dengue Hemorrhagic Fever; Flavivirus
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Biological Products; Vaccines; Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- TDENV-PIV alum4 (Experimental): 4 µg TDENV-PIV with Alum adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Biological: Biological/Vaccine: 4 µg TDENV-PIV with Alum adjuvant
- TDENV-PIV AS03B (Experimental): 1 µg TDENV-PIV with AS03B adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Biological: Biological/Vaccine: 1 µg TDENV-PIV with AS03B adjuvant
- Placebo (Placebo Comparator): Phosphate buffered saline; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Other: Phosphate buffered saline
- TDENV-PIV alum1 (Experimental): 1 µg TDENV-PIV with Alum adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Biological: 1 µg TDENV-PIV with Alum adjuvant
- TDENV-PIV AS01E (Experimental): 1 µg TDENV-PIV with AS01E adjuvant; 0.5 mL intramuscular injection at 0 and 28 days
  Interventions: Biological: 1 µg TDENV-PIV with AS01E adjuvant

INTERVENTIONS:
Biological: Biological/Vaccine: 4 µg TDENV-PIV with Alum adjuvant
  Arms: TDENV-PIV alum4
Biological: Biological/Vaccine: 1 µg TDENV-PIV with AS03B adjuvant
  Arms: TDENV-PIV AS03B
Other: Phosphate buffered saline
  Arms: Placebo
Biological: 1 µg TDENV-PIV with Alum adjuvant
  Arms: TDENV-PIV alum1
Biological: 1 µg TDENV-PIV with AS01E adjuvant
  Arms: TDENV-PIV AS01E

SUMMARY:
This is a first time in humans (FTiH) study designed to assess the experimental TDENV-PIV vaccine in a predominantly dengue-primed adult population. The study is designed to afford a first time in humans (FTiH) safety and immunogenicity assessment of three TDENV-PIV vaccine candidates, each formulated with a different adjuvant: either aluminum hydroxide, AS01E or AS03B (adjuvants used in GSK Biologicals' hepatitis B candidate vaccine, malaria candidate vaccine and pandemic flu vaccine, respectively). Each vaccine candidate will contain 1 µg of purified virus antigen per each of the four DENV types. Additionally, the study will evaluate an alum adjuvanted TDENV-PIV vaccine candidate containing 4 µg of purified virus antigen per each of the four DENV types. The control group will receive a saline placebo. All experimental vaccinations will be administered according to a 2-dose schedule, 28 days apart. There is a parallel FTiH study that is conducted in the United States in a dengue-naive population using the same investigational vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits, etc.)
* A male or female between 20 and 39 years of age (inclusive) at the time of consent
* Written informed consent obtained from the subject
* Healthy subjects as established by medical history and clinical examination before entering into the study
* Subject has lived in the Caribbean for more than 10 years
* Female subjects of non-childbearing potential (non-childbearing potential is defined as having either a current tubal ligation at least three months prior to enrollment, hysterectomy, ovariectomy, or is post-menopause).
* Female subjects of childbearing potential may be enrolled in the study, if the subject has:

  * practiced adequate contraception for 30 days prior to vaccination, and
  * a negative urine pregnancy test on the day of vaccination, and
  * agreed to continue adequate contraception until two months after completion of the vaccination series

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines/placebo during the period starting 30 days preceding the first dose of study vaccine/placebo and/or planned use during the study period
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 180 days prior to the first vaccine/placebo dose (for corticosteroids, this will mean prednisone ≥ 20 mg/day or equivalent; inhaled and topical steroids are allowed)
* Planned administration or administration of a vaccine/product not foreseen by the study protocol during the Exclusion:
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines/placebo during the period starting 30 days preceding the first dose of study vaccine/placebo and/or planned use during the study period
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 180 days prior to the first vaccine/placebo dose (for corticosteroids, this will mean prednisone ≥ 20 mg/day or equivalent; inhaled and topical steroids are allowed)
* Planned administration or administration of a vaccine/product not foreseen by the study protocol during the period starting 30 days prior to the first dose of vaccine/placebo until after the visit at Day 56 (if influenza activity warrants vaccination of healthy young adults, influenza vaccination will be encouraged and will not lead to study exclusion)
* Previous or planned administration of any other flavivirus vaccine (approved or investigational) for the entire study duration
* Previous receipt of any investigational dengue virus vaccine
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency
* History of, or current auto-immune disease
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine/placebo or related to a study procedure
* Major congenital defects or serious chronic illness
* History of any neurological disorders or seizures
* Acute disease and/or fever (≥37.5°C/99.5°F oral body temperature) at the time of enrollment (a subject with a minor illness, i.e., mild diarrhea, mild upper respiratory infection, etc., without fever, may be enrolled at the discretion of the investigator)
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
* Administration of immunoglobulins and/or any blood products during the period starting 90 days preceding the first dose of study vaccine/placebo or planned administration during the study period
* History of chronic alcohol consumption and/or drug abuse
* Pregnant or lactating female or female planning to become pregnant or planning to discontinue contraceptive precautions
* A planned move to a location that will prohibit participating in the trial until study end for the participant
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* Subject seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV)
* Safety laboratory test results that are outside the normal limits for their age, gender, and locality at screening.

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Safety and reactogenicity of various TDENV-PIV formulations from Day 0 through 28 days after the second dose (Day 0 - Day 56) | Up to Day 56
  Safety and Reactogenicity:
  * Occurrence, intensity and relationship to vaccination of solicited local and general adverse events (AEs) during the 7-day follow-up period post each vaccination (Day 0-6)
  * Occurrence, intensity and relationship to vaccination of unsolicited AEs during the 28-day follow-up period post each vaccination (Day 0-27)
  * Hematological and biochemical levels at study visits on Days 0, 7, 28, 35 and 56
  * Occurrence of serious adverse events (SAEs) from Day 0 to Day 56
  * Occurrence of potential immune-mediated diseases (pIMDs) and medically attended AEs from Day 0 to Day 56
Humoral immunogenicity to each of four DENV types of various TDENV-PIV formulations 28 days after the second dose (Day 56) | Day 56
  Humoral Immunogenicity:
  Neutralizing antibody titers specific to each DENV type at Day 56
  * Geometric mean titers (GMTs) of neutralizing antibody titers to each DENV type
  * Rate of fold increases in neutralizing antibody from Day 0 for each DENV type
  * Seropositivity rates for each DENV type
  * Trivalent and tetravalent seropositivity rates

SECONDARY OUTCOMES:
Safety of various TDENV-PIV formulations, from Day 0 to Month 13 (Visits 1-11) | Up to month 13
  Safety:
  * Hematological and biochemical levels at study visits on Months 4, 7, 10 and Month 13
  * Occurrence of pIMDs and medically attended AEs from Day 0 to Month 13
  * Occurrence of any SAE from Day 0 to Month 13
Humoral immunogenicity to each of four DENV types of various TDENV-PIV formulations on Days 0, 7 and 28 and Months 7 and 13 | Up to month 13
  Humoral Immunogenicity:
  * Geometric mean titers (GMTs) of neutralizing antibody titers to each DENV type
  * Rate of fold increases in neutralizing antibody from Day 0 for each DENV type
  * Seropositivity rates for each DENV type
  * Trivalent and tetravalent seropositivity rates
• To evaluate the safety of various TDENV-PIV formulations from Month 14 through the end of the study (Visit 15) | Up to the end of study (Month 37-39)
  Occurrence of serious adverse events (SAEs) related to study procedures from Month 14 to end of study (Month 37-39)

CONTACTS AND LOCATIONS:
Overall Officials: Clemente Diaz, MD, Principal Investigator — University of Puerto Rico
Locations (1):
- Clinical Research Center, 1st Floor University Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Diaz C, Lin L, Martinez LJ, Eckels KH, Campos M, Jarman RG, De La Barrera R, Lepine E, Toussaint JF, Febo I, Innis BL, Thomas SJ, Schmidt AC. Phase I Randomized Study of a Tetravalent Dengue Purified Inactivated Vaccine in Healthy Adults from Puerto Rico. Am J Trop Med Hyg. 2018 May;98(5):1435-1443. doi: 10.4269/ajtmh.17-0627. Epub 2018 Mar 1. PMID 29512481